CLINICAL TRIAL: NCT05170386
Title: Effect of Cognitive Training on Sleeping Disorders in Stroke: a Randomized Controlled Trial
Brief Title: Cognitive Training on Sleeping Disorders in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Lama Saad El-Din Mahmoud, Lecturer of physical therapy, Department of Neuromuscular disorders and its surgery, faculty of physical therapy, october 6 univerisity, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T. REC/012/003445
Record Dates: First submitted 2021-12-10; First posted 2021-12-28 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Sleep Disorder
Keywords: Stroke; sleep disorders; cognition
MeSH Terms: conditions — Stroke; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: group A (20 patients): that will receive cognitive training combined with instructive conventional treatment for sleeping disorder, and group B (20 patients): that will receive instructive conventional treatment for sleeping disorder
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): receive cognitive training combined with instructive conventional treatment for sleeping disorder
  Interventions: Other: Cognitive training Therapy; Other: instructive conventional treatment
- control group (Experimental): receive instructive conventional treatment for sleeping disorder
  Interventions: Other: instructive conventional treatment

INTERVENTIONS:
Other: Cognitive training Therapy — Cognitive training Therapy include: Writing the reminiscences
  • Solving a table• Writing a letter making a calendar and writing a note about the daily activities on it Facing patients' fears instead of avoiding them.Using role-playing to prepare for potentially problematic interactions with others.Learning to calm one's mind and relax one's body.
  Arms: study group
Other: instructive conventional treatment — instructive conventional treatment breathing relaxation exercise inform of diaphragmatic breathing Practice sleep hygiene such as keeping a regular sleep schedule. Get regular exercise. Minimize noise. Minimize light. Manage the temperature so that you're comfortable.

SUMMARY:
Cognitive impairment and sleeping disturbance following stroke diagnosis are common symptoms that significantly affect the quality of life.

DETAILED DESCRIPTION:
40 patients from both sexes will participate in this study. All the patients have to be diagnosed as stroke patients. The patients will be divided into two groups; group A (20 patients): which will receive cognitive training combined with instructive conventional treatment for a sleeping disorder, and group B (20 patients): which will receive instructive conventional treatment for sleeping disorder all the patients will be assessed pre and post-treatment using 1- Epworth sleeping scale, 2-Pittsburgh sleep quality index ( PSQI) 3- MINI mental cognitive scale

ELIGIBILITY:
Inclusion Criteria:

* stroke onset at least 5 months prior to study enrolment
* with sleeping disturbance
* age will range from 40:55
* upper extremity spasticity ranging from
* according to Modified Ashowrth Scale.

Exclusion Criteria:

* difficulty to communicate
* other neurological conditions that cause sleeping disorders
* severe depression or other psychiatric symptoms.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Epworth sleeping scale (ESS) | 4 weeks
  The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. Most people engage in those activities at least occasionally, although not necessarily every day. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'. The questionnaire takes no more than 2 or 3 minutes to answer. It is available in many different languages.
Pittsburgh sleep quality index ( PSQI) | 4 weeks
  0 self-reported items Minimum score: o; Maximum score: 21 0-3 scoring for each of the 7 components Higher scores indicate worse sleep quality
  • 7 components/sub-scales: subjective sleep qualitv, sleep latenev, sleep duration.
  habitual sleep efficiency, sleep disturbances, use of sleeping medications and daytime dysfunction

SECONDARY OUTCOMES:
The Mini-Mental State Examination (MMSE) | four weeks
  The Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairmen Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment

CONTACTS AND LOCATIONS:
Locations (1):
- Lama S Mahmoud, Al Jīzah, Select State, Egypt

IPD SHARING:
Plan to Share IPD: No